CLINICAL TRIAL: NCT00874536
Title: The Effect of Omega-3 Fatty Acid Supplementation on Behavior of Children With ADHD
Brief Title: Omega-3 Supplementation and Attention-deficit-hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Israel Association of Pediatricians (Unknown)
Responsible Party: Principal Investigator, gal dubnov raz, Senior physician, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDR3-HMO-CTIL
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; methylphenidate; omega-3
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALA (Experimental): This group will receive the ALA supplement
  Interventions: Dietary Supplement: omega-3 fatty acid alpha-linolenic acid (ALA)
- Placebo (Placebo Comparator): This group will receive the placebo supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid alpha-linolenic acid (ALA) — 3 grams of ALA-containing plant oil
  Arms: ALA
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
It is assumed that only 1/5 of children diagnosed with attention-deficit-hyperactivity disorder (ADHD) are treated. New treatment modalities are urgently needed. Omega-3 fatty acids have been used in this setting, yet results are conflicting. The parent omega-3 fatty acid alpha-linolenic acid (ALA) has only been used in one trial. 40 children diagnosed with ADHD will be randomized to consume either ALA or placebo for two months. Baseline and end assessments will include ADHD-related questionnaires and a computerized test. The investigators hypothesize that ALA supplementation will prove beneficial for children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* informed consent

Exclusion Criteria:

* refusal of any testing
* any comorbidities
* any medication or supplement use

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms | 8 weeks
  scores of DSM and Conners questionnaires

SECONDARY OUTCOMES:
Computerized test performance | 8 weeks
  performance in a computerized test of attention

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Jerusalem, Israel

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600